CLINICAL TRIAL: NCT03008148
Title: Randomized Phase II/III Trial of Radiotherapy Plus Concomitant and Adjuvant Temozolomide With or Without Hydroxychloroquine, Rapamycin for Newly Diagnosed Glioblastoma
Brief Title: Phase II/III Trial of CCRT With or Without JP001 for Newly Diagnosed GBM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johnpro Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP001-GM-001
Record Dates: First submitted 2016-12-23; First posted 2017-01-02 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiation,Temozolomide (Active Comparator): 1. CCRT Phase: Radiation(60 Gy in 2 Gy/fx) + daily Temozolomide (75 mg/m²/day for 6 weeks).
  2. Rest Phase: Rest for 4 weeks.
  3. Chemotherapy Phase: Temozolomide 150-200 mg/m² Day 1-5 of 28-Day for a maximum of 6 cycles.
  4. Maintenance Phase: No maintenance treatment until disease progression confirmed.
  Interventions: Radiation: CCRT; Drug: Temozolomide
- Radiation,Temozolomide,Siroquine(JP001) (Experimental): 1. CCRT Phase: Radiation(60 Gy in 2 Gy/fx) + daily Temozolomide (75 mg/m²/day for 6 weeks) + Daily JP001 (2 tablets once a day for 6 weeks).
  2. Rest Phase: Daily JP001(2 tablets/day) for 4 weeks.
  3. Chemotherapy Phase: Temozolomide 150-200 mg/m² Day 1-5 of 28-Day for a maximum of 6 cycles + Daily JP001(2 tablets once a day) for 24 weeks (4 weeks for each cycle).
  4. Maintenance Phase: JP001(2 tablets once a day) until disease progression confirmed.
  Interventions: Radiation: CCRT; Drug: Temozolomide; Drug: Siroquine

INTERVENTIONS:
Radiation: CCRT — CCRT Phase: Radiation(60 Gy in 2 Gy/fx) + daily Temozolomide (75 mg/m²/day for 6 weeks).
Drug: Temozolomide — Temozolomide 150-200 mg/m² Day 1-5 of 28-Day for a maximum of 6 cycles.
  Other Names: Chemotherapy
Drug: Siroquine — 1. Chemotherapy Phase: Temozolomide 150-200 mg/m² Day 1-5 of 28-Day for a maximum of 6 cycles + Daily JP001(2 tablets once a day) for 24 weeks (4 weeks for each cycle).
  2. Maintenance Phase: JP001(2 tablets once a day) until disease progression confirmed.
  Other Names: JP001
  Arms: Radiation,Temozolomide,Siroquine(JP001)

SUMMARY:
This is a multi-center, phase II/III, open-label, randomized, parallel and standard chemoradiation-controlled study where eligible subjects will be randomized at 1:1 ratio to receive control treatment or study treatment. The primary objective of this trial is to evaluate the effect of add-on JP001 to standard chemoradiation in increasing overall survival (OS) on newly diagnosed glioblastoma (GBM) patients.

DETAILED DESCRIPTION:
After enrollment, subjects' previous tumor block used for glioblastoma diagnosis that is consented to provide during the study period will be sent to a central laboratory for the assessment of MGMT status. Moreover, subjects will be randomized in either Control or Study arm at Visit 2. Subjects in Control arm will receive a standard chemoradiation. However, subjects in Study arm will receive a standard chemoradiation in combination with concurrent JP001 in whole study period. During the study, a sufficient amount of investigational products will be supplied to subjects in study groups until next scheduled visits. Subjects will self-administer investigational product orally with water at approximately the same time in each day. Subjects should fast for a minimum of 2 hours prior to any doses of JP001 and/or Temozolomide and then fast for another 1 hour after taking JP001 and/or Temozolomide. During and at the end of treatment, subjects will be evaluated for efficacy and safety parameters. Moreover, there will be a Follow-up visit for safety 4 weeks after the End-of-Treatment visit. If a subject is early withdrawn from the study, the End-of-Treatment visit should be arranged and all assessments assigned in this visit should be performed. The Safety Follow-up visit for early withdrawn subjects could be either clinic visit or telephone contact. If withdrawn subjects refuse to perform Follow-up visit, the Follow-up visit is allowed to cancel. For subjects who completed or discontinued study treatment, assessment of survival status will be performed every 8 weeks by telephone contact until death, study end (last subject last visit; the last subject needs to be followed at least 30 months), or study termination by Sponsor. Survival information will be recorded in the medical source and CRF. If subjects are lost to follow-up or refuse to receive the assessment of survival status, the investigator will record the last date subjects known to be alive in the medical source and case report form.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically proven newly diagnosed case of GBM (WHO grade IV) and treatment-naive (chemotherapy and radiotherapy) for GBM. Diagnosis must be made by stereotactic biopsy or surgical excision, either partial or complete within 3 months prior to Visit 1.
2. Subject's RPA class is class III, IV or V.
3. Subjects with stereotactic biopsy or brain surgery must be suited for or will be scheduled for CCRT followed by Temozolomide treatment, the standard treatment recommended by institutes and fulfilled the reimbursement guideline of National Health Insurance Administration.
4. Subjects must have recovered from the effects of surgery, post-operative infection, and other complications prior to Visit 1. Study treatment must be performed > 3 weeks and ≤ 8 weeks after craniotomy. Ventricular fluid reservoir or Ventriculo-Peritoneal shunting tube is allowed to keep.
5. A diagnostic contrast-enhanced MRI of the brain must be performed postoperatively within 28 days prior to Visit 2 (Day 1).
6. ECOG performance status ≤ 3 at Visit 1.
7. Age from 20 to 80 years old at Visit 1.
8. Life expectation ≥ 12 weeks at Visit 1.
9. CBC/differential obtained at Visit 1, with adequate bone marrow function defined as follows:

   1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 (1.5 x 109/L) or white blood cell (WBC) ≥ 3,000 cells/mm3 (3 x 109/L).
   2. Platelets count ≥ 100,000 cells/mm3 (100 x 109/L).
   3. Hemoglobin (Hgb or Hb) ≥ 10.0 g/dL (100 g/L) (Note: The use of transfusion or other intervention to achieve Hemoglobin ≥ 10.0 g/dL (100 g/L) is acceptable).
10. Adequate renal function, as defined below:

    a. Creatinine ≤ 1.5 times upper laboratory limit at Visit 1.
11. Adequate hepatic function, as defined below:

    1. Total Bilirubin ≤ 2.0 mg/dL (34.20 umol/L) at Visit 1.
    2. ALT ≤ 3 times upper laboratory limit at Visit 1.
    3. AST ≤ 3 times upper laboratory limit at Visit 1.
12. Subjects is able to understand and willing to comply with the study procedures and has signed the informed consent form (ICF).

Exclusion Criteria:

1. Other invasive malignancy. However, subject with other invasive malignancy that have been disease-free more than or equal to 10 years and deemed no need for anti-cancer treatments can be recruited. Subjects with noninvasive malignancy, including carcinoma in situ of the breast, non-melanomatous skin cancer and cervix carcinoma in situ can be recruited if disease-free and treatment free more than or equal to 3 years.
2. Metastases detected beyond the cranial vault.
3. Subjects with the following history:

   1. Brain irradiation or Temozolomide usage.
   2. Macular degeneration or retinopathy.
   3. Renal transplantation.
4. Subjects are currently receiving any anti-rejection medicine or Hydroxychloroquine sulfate for rheumatoid arthritis.
5. Subjects with severe and active co-morbidity, defined as follows:

   1. Clinical active kidney, liver, lung or cardiac disease.
   2. Acute bacterial or fungal infection requiring intravenous antibiotics at Visit 1 and acquired immune deficiency syndrome (AIDS).
   3. Any active infection or uncontrolled infection at Visit 1.
   4. Abnormal CXR finding with risks of infection and interstitial lung disease/pneumonitis.
6. Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant from study drug.
7. Mean QTc > 500 msec (with Bazett's correction), history of familial long QT syndrome or other significant ECG abnormality noted at Visit 1.
8. Known hypersensitivity reactions to Temozolomide, dacarbazine (DTIC), hydroxychloroquine, 4-aminoquinoline, rapamune, sirolimus, rapamycin, or their analogs.
9. Women of child-bearing potential or men who are able to father a child unwilling to use a. medically acceptable method of contraception during the trial.
10. Subjects participated in another investigational agent study in the past 30 days or are planning to do so during the study period.
11. Subjects are considered ineligible for the study as judged by the investigator.
12. Subjects with positive HBsAg or positive anti-HCV.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival time. | 120 weeks
  All subjects will be followed until study end (the date of last subject last visit; the last subject need to be followed at least 30 months) or death, whichever comes first; OS defined as the time from the date of Randomization to the date of death or last follow-up.

SECONDARY OUTCOMES:
Progression-free survival time | 120 weeks
  All subjects will be followed until study end or disease progression confirmed, whichever comes first; PFS defined as the time from the date of Randomization to the date of disease progression, death or last follow-up.
OS rate at 1 year. | 1 year
  OS defined as the time from the date of Randomization to the date of death or last follow-up.
PFS rate at 1 year. | 1 year
  PFS defined as the time from the date of Randomization to the date of disease progression, death or last follow-up.
The time and rate of OS in different RPA class. | 120 weeks
The time and rate of PFS in different RPA class. | 120 weeks
Objective response rate. | 120 weeks
  Defined as the proportion of subjects who were confirmed completed response or partial response determined by RANO criteria.
Changes in score of EORTC QLQ-C30 | 120 weeks
Changes in score of EORTC QLQ-BN20. | 120 weeks
Changes in grade of ECOG performance status. | 120 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No